CLINICAL TRIAL: NCT01912521
Title: Mfangano Island Healthy Networks Impact Study
Acronym: MIHNIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Organic Health Response (Other); Microclinic International (Other); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIHNIS
Record Dates: First submitted 2013-07-23; First posted 2013-07-31 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: HIV
Keywords: HIV; Stigma; Social support; Social network; Kenya
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): This arm is eligible for participation in the Mfangano Health Net Microclinic Program, a social network-based educational program.
  Interventions: Behavioral: Mfangano Health Net Microclinic Program
- Comparison (No Intervention): This arm is not eligible for participation in the intervention. Participants still have access to usual care at the Sena Health Center or their health facility of choice.

INTERVENTIONS:
Behavioral: Mfangano Health Net Microclinic Program — Educational program in which HIV positive individuals are invited to recruit their social networks to form 'microclinic' groups. These groups participate in a 6-month educational curriculum composed of information on HIV biology, interpersonal communication strategies and community mobilization. At the conclusion of the program, participants are encouraged to disclose their HIV status to members of their group through a facilitated disclosure process.
  Arms: Intervention

SUMMARY:
This pilot study is a non-randomized controlled cohort study evaluating the impact of social network-based HIV education on antiretroviral therapy (ART) adherence, clinical outcomes, food security, social support, HIV knowledge, and risk behaviors among people living with HIV/AIDS, as well as members of their associated social support networks. The intervention, known as the Mfangano Health Net Microclinic Pilot Program, consists of a 6-month education program on HIV biology, interpersonal communication and community mobilization for both HIV positive individuals and their self-selected social network members selected irrespective of HIV status. Investigators hypothesize that participation in the microclinic program will improve ART adherence, cluster of differentiation 4 (CD4) count, social support, HIV knowledge and food insecurity and will reduce HIV-related stigma, as compared to participants in control communities.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive patient on ART at Sena Health Center or member of patient's social network
* Resident of Mfangano Island
* 18 years of age or older
* conversant in DhoLuo or English languages

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 883 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Antiretroviral therapy (ART) Adherence | change from baseline to 6-months
  change in ART drug levels measured in small hair samples from baseline to 6 months
Disengagement from care | From time of study enrollment to first instance of 90-day gap in care, censorship (death, transfer outside study area) or end of study (up to 22 months)
  Incidence of missing a clinic appointment by ≥90 days without having first transferred care to another clinic or died.

SECONDARY OUTCOMES:
Stigma | change from baseline to 6-months
  stigma as measured by Parallel HIV/AIDS Stigma Scale (Attributed Stigma Attitudes)
Social support | change from baseline to 6-months
  Social support as measured by Duke-University of North Carolina (UNC) Functional Social Support Scale
HIV knowledge | change from baseline to 6-months
  HIV knowledge as measured by HIV Knowledge Questionnaire ("HIV-KQ-18")
Time in care | From time of study enrollment until study closure (22 months) or censorship (death or transfer of care to facility outside study area)
  Proportion of time eligible for HIV care that patient is adherent to clinic appointment schedules. Calculated by subtracting the sum of all gaps in care from the total time eligible for care, and dividing by total time eligible for care. Gaps in care are defined as the number of days between a missed appointment and subsequent return to any clinic in the study area to access HIV care.
ART adherence - end of study | change from baseline to end of study (22 months)
  change in ART drug levels measured in small hair samples from baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Cohen, MD, Principal Investigator — University of California, San Francisco; Elizabeth Bukusi, MBChB, M.Med, Principal Investigator — Kenya Medical Research Institute; Charles R Salmen, MSc, MD Candidate, Principal Investigator — University of California, San Francisco; Matthew D Hickey, MD Candidate, Principal Investigator — University of California, San Francisco
Locations (1):
- Ekialo Kiona Center, Kitawi Beach, Mfangano Island, Nyanza, Kenya